CLINICAL TRIAL: NCT05062993
Title: Evaluation of the Effect of Ultrasound Guided Caudal Epidural Pulsed Radiofrequency Stimulation on Chronic Pain in Patients With Failed Back Surgery Syndrome
Brief Title: Evaluation of the Effect of Caudal Epidural Pulsed Radiofrequency Stimulation on Chronic Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Diskapi Teaching and Research Hospital (Other)
Responsible Party: Principal Investigator, Selin Guven Kose, Principal Investigator, Diskapi Teaching and Research Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 98/08
Record Dates: First submitted 2021-07-07; First posted 2021-09-30 (Actual); Last update posted 2022-02-07 (Actual); Status verified 2022-01

CONDITIONS: Pain, Chronic
Keywords: caudal epidural stimulation; chronic pain; lumbosacral radiculopathy; postlumbar surgery syndrome
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- study group (Experimental): Patients with chronic radicular pain will be included in this study. Ultrasound guided caudal epidural pulse radiofrequency technique will be applied to the study group.
  Interventions: Procedure: caudal epidural pulse radio frequency

INTERVENTIONS:
Procedure: caudal epidural pulse radio frequency — A needle is inserted into the caudal epidural space under ultrasound guidance and pulse radiofrequency is administered at 5 Hz using a 5. ms pulse width for 600 seconds at 55 V.

SUMMARY:
Postlumbar surgery syndrome (PLSS; failed back syndrome) is characterized by persistent pain in the lower back or lower extremities after spinal surgery. It occurs in 10-40% of patients who undergo a back surgery. The recently introduced pulsed radiofrequency (PRF) technique is widely used to provide relief from chronic pain and studies have shown that PRF stimulation can be used to control neuropathic pain by placing the needle electrodes into the caudal epidural space The aim of this study is evaluation of the effect of ultrasound guided caudal epidural pulsed radiofrequency stimulation in patients with chronic lumbosacral radicular pain due to postlumbar surgery syndrome.

ELIGIBILITY:
Inclusion Criteria:

* chronic pain in legs or back pain
* unsatisfactory response to at least one transforaminal, lumbar or caudal steroid injections

Exclusion Criteria:

* coagulation disorders
* psychiatric disorders
* rheumatoid disorders
* infections

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-02-22 (Actual); Primary Completion 2021-05-01 (Actual); Study Completion 2021-07-01 (Actual)

PRIMARY OUTCOMES:
Numeric Rating Scale(NRS) (0-10) | before procedure
  The 11-point NRS consists of numbers between 0 and 10 where 0 indicates "no pain" and 10 indicates "maximum pain." The patient is instructed to identify one number between 0 and 10, which is best representative of their pain intensity.
Numeric Rating Scale | 2 weeks after procedure
  The 11-point NRS consists of numbers between 0 and 10 where 0 indicates "no pain" and 10 indicates "maximum pain." The patient is instructed to identify one number between 0 and 10, which is best representative of their pain intensity.
Numeric Rating Scale | 4 weeks after procedure
  The 11-point NRS consists of numbers between 0 and 10 where 0 indicates "no pain" and 10 indicates "maximum pain." The patient is instructed to identify one number between 0 and 10, which is best representative of their pain intensity.
Numeric Rating Scale | 8 weeks after procedure
  The 11-point NRS consists of numbers between 0 and 10 where 0 indicates "no pain" and 10 indicates "maximum pain." The patient is instructed to identify one number between 0 and 10, which is best representative of their pain intensity.

CONTACTS AND LOCATIONS:
Overall Officials: Selin Guven Kose, Principal Investigator — Diskapi Yildirim Beyazit Education and Research Hospital
Locations (1):
- Diskapi Yildirim Beyazit Training and Research Hospital, Ankara, Turkey (Türkiye)